CLINICAL TRIAL: NCT05004376
Title: Text-based Intervention to Improve Adherence to Colorectal Cancer Screening Recommendations Among Emergency Department Patients
Brief Title: Text-based Colorectal Cancer Prevention Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Beau Abar, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 00006479
Record Dates: First submitted 2021-07-28; First posted 2021-08-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with a prospectively collected convenience sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-adherent control (No Intervention): Control subjects will receive no text intervention and a 150 day follow-up phone call.
- Non-adherent intervention (Experimental): Intervention subjects will receive the text messaging intervention and a 150 day follow-up phone call.
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Text Messaging — Text messages based on behavioral theory to encourage scheduling colorectal cancer screening.
  Arms: Non-adherent intervention

SUMMARY:
In this project, we intend to conduct a randomized pilot trial of a structured behavioral intervention, grounded in the Theory of Planned Behavior and Self-Determination Theory, to promote adherence of patients aged 45 - 75 to USPSTF colorectal cancer screening recommendations. We will also collect qualitative feedback on perceptions of the intervention to inform its refinement.

DETAILED DESCRIPTION:
The investigators propose a pilot randomized controlled trial with a prospectively collected convenience sample of 130 ED patients non-adherent with CRC screening guidelines over a 3-month period. ED Research Associates (EDRAs) will use the EPIC eRecord system to screen adult patients registered in the ED at URMC and Noyes Memorial Hospital (when an EDRA is present in that ED) for eligibility. Inclusion criteria will include: 45-75 years and English or Spanish speaking (costs for interpreting study surveys and patient interactions will be paid for from PI discretionary research funds). Exclusion criteria will include personal and/or family history of colorectal cancer, personal history of inflammatory bowel disease, and a history of abdominal or pelvic radiation to treat a prior cancer. These exclusions were chosen due to their impact on standard colorectal screening recommendations. After consent, subjects will complete a ~10-minute questionnaire administered by the EDRA to determine adherence to current USPSTF guidelines for colorectal cancer screening using validated items in the CDC's National Health Interview Survey16. The enrollment process will categorize study participants into three groups: adherent, uncertain, or non-adherent. Subjects found to be adherent will be notified and their participation will conclude. Subjects found to be in the uncertain or non-adherent groups will be randomized into the treatment or control condition. Following intervention, subjects who were non-adherent will be referred to their usual care provider to discuss options for becoming adherent. Subjects for whom adherence is uncertain will be referred to their usual care provider to confirm their adherence status. Subjects who find through their PCP that they are adherent will be treated as screen failures. Sensitivity analyses will be performed to evaluate estimates of intervention efficacy with and without inclusion of subjects initially determined uncertain and later categorized as non-adherent. Following the initial enrollment, randomization, and recommendation to contact their PCPs, subjects in the intervention condition will receive a series of 6 text messages, sent at approximately 15 day intervals, presenting theory-based messages aimed at encouraging colorectal cancer screening uptake. Subjects without a primary care provider will be given information on how to establish a PCP in Rochester and on cancer screening services subsidized through the Cancer Services Program (CSP) of the Finger Lakes Region (our current R01 includes referrals to the CSP). All subjects in the non-adherent and uncertain groups will receive a follow-up call at 150 days for a ~5-minute survey to determine if they underwent or scheduled screening, if they learned that they did not require screening, and what barriers they perceived in getting screened. Qualitative feedback regarding perceptions of the intervention will also be collected in order to refine the intervention for future study. Medical chart review will also be conducted to confirm patient self-reports, making use of UR records and records from the Rochester Regional Health Information Organization (RHIO; our current R01 has incorporated the RHIO).Completion of a "second-level" consent form for use of the RHIO for chart review will be required for enrollment. In our cervical cancer pilot study, we successfully contacted 68% of participants for follow-up, 11 of whom declined to complete the follow-up interview. Based on lessons learned in our preliminary work, we have developed several strategies (currently employed in our R01 study), in addition to the incentive payment for study completion, which we will employ to maximize retention in this study:

1. Telephone numbers will be confirmed in the ED during enrollment by the EDRA performing the enrollment by calling the patient's phone to be certain the number is correct.
2. Up to five calls will be made to each study participant during the follow-up window.
3. Each participant will be provided with study team contact information and asked to notify us in the event that their phone number changes.
4. In addition to their primary cell phone number, alternative contact information will be sought from each participant to enable attempts at re-engagement, including: a.Secondary telephone number of participant b.Email address(es) and mailing address.
5. The EHR will be accessed to check for changes in contact information

ELIGIBILITY:
Inclusion Criteria:

* Present at Strong Memorial Hospital or Noyes Community Hospital Emergency Departments
* Age 45-75
* English or Spanish speaking
* Capacity to consent

Exclusion Criteria:

* Personal and/or family history of colorectal cancer
* Personal history of inflammatory bowel disease
* History of abdominal or pelvic radiation to treat a prior cancer
* Non-English and Non-Spanish speaking
* Inability to consent
* Lack of text-capable mobile phone and/or inability to use text function

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Screening | 150 days
  Rates of completed or scheduled screening

SECONDARY OUTCOMES:
Phone Interview for refinement of Intervention | 150 days
  Collect qualitative feedback on perceptions of the intervention to inform its refinement.

CONTACTS AND LOCATIONS:
Locations (1):
- Strong Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abar B, Park CS, Wood N, Marino D, Fiscella K, Adler D. Intervention to increase colorectal cancer screening among emergency department patients: results from a randomised pilot study. Emerg Med J. 2024 Jun 20;41(7):422-428. doi: 10.1136/emermed-2023-213761. PMID 38777559